CLINICAL TRIAL: NCT00154180
Title: Effects of Estrogen Replacement on Atherosclerosis Progression in Recently Menopausal Women
Brief Title: Kronos Early Estrogen Prevention Study (KEEPS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kronos Longevity Research Institute (Other)
Collaborators: Albert Einstein College of Medicine (Other); Brigham and Women's Hospital (Other); Columbia University (Other); Mayo Clinic (Other); University of California, San Francisco (Other); University of Utah (Other); University of Washington (Other); Yale University (Other)
Responsible Party: S. Mitchell Harman, MD, PhD/Director, Kronos Longevity Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KLRI-04-1; WIRB Protocol #20040792; NCT00623311 (obsolete NCT alias)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Menopause; Arteriosclerosis
Keywords: Perimenopause; Coronary Disease; Estrogen Replacement Therapy; Hormone Replacement Therapy
MeSH Terms: conditions — Arteriosclerosis; Coronary Disease | interventions — Estrogens, Conjugated (USP); Estradiol; Progesterone; 2-chloroethyl ethyl sulfide; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): CEE 0.45 mg w/ Prometrium 200 mg patch 0.05 mg w/ Prometrium 200 mg
  Interventions: Drug: Conjugated equine estrogens 0.45 mg/day; Drug: Transdermal estradiol, 50 mcg/day; Drug: Micronized progesterone, 200 mg/day x 12 d/month; Drug: CEE, progesterone, transdermal patch or the placebo
- Arm 2 (Placebo Comparator): Placebo patch, placebo CEE, placebo Prometrium
  Interventions: Drug: CEE , progesterone, estradiol patch or placebo for each; Drug: CEE, progesterone, transdermal patch or the placebo

INTERVENTIONS:
Drug: Conjugated equine estrogens 0.45 mg/day — Pill, 1 pill taken daily each month for the study duration
  Other Names: Premarin or placebo
  Arms: Arm 1
Drug: Transdermal estradiol, 50 mcg/day — Patch; 1 patch is applied to the skin weekly. Patch site is rotated on a weekly basis.
  Other Names: Climara 50 mcg/day or placebo
  Arms: Arm 1
Drug: Micronized progesterone, 200 mg/day x 12 d/month — capsule, 1 capsule taken daily for the first 12 days of each month for the study duration
  Other Names: Prometrium or placebo
  Arms: Arm 1
Drug: CEE , progesterone, estradiol patch or placebo for each — CEE 0.45mg 1 PO QD Progesterone 200 mg 1 PO HS first 12 days of the month estradiol patch use 1 per week
  Other Names: Premarin; Prometrium; Climara Patch
  Arms: Arm 2
Drug: CEE, progesterone, transdermal patch or the placebo — CEE 0.45 mg 1 PO QD or placebo equivalent Prometrium 200 mg 1 PO qHS for first 12 dasy of each month or placebo equivalent transdermal patch 0.05 mg use 1 patch per week or placebo equivalent
  Other Names: Premarin; Prometrium; Climara

SUMMARY:
The study will examine the effects of estrogen and progesterone on the development of atherosclerosis in menopausal women when hormone treatment is initiated within 3 years of the menopausal transition.

DETAILED DESCRIPTION:
The KEEPS is designed to explore the hypothesis that early initiation of hormone therapy, in women who are at the inception of their menopause, will decrease the rate of accumulation of atherosclerotic plaque, indicating a likely delay in the onset of clinical cardiovascular disease. The study is designed as a multicenter, 4 year randomized clinical trial. It will evaluate the effectiveness of of 0.45 mg/day of oral conjugated equine estrogens or 50 mcg/day of transdermal estradiol via skin patch changed weekly (each in combination with cyclic oral, micronized progesterone, 200 mg daily for 12 days per month), versus placebo in preventing progression of carotid intimal medial thickness by sonogram and the accrual of coronary calcium in women aged 42-58 who are within 36 months of their final menstrual period at initiation of treatment. A number of secondary endpoints including biochemical and genetic risk factors for cardiovascular and thrombotic disease, and effects on cognition will also be studied. The study will enroll a total of 720 women in 2005-6, with an anticipated completion of the trial in 2010.

ELIGIBILITY:
Inclusion Criteria:

* menses absent for at least 6 months and no more than 36 months
* good general health
* plasma FSH level greater than or equal to 35 mIU/ml
* estradiol levels < 40 pg/ml
* normal mammogram within 1 year of randomization

Exclusion Criteria:

* use of hormone replacement or supplement within 3 months of randomization
* endometrial thickness >5 mm by vaginal ultrasound
* in utero exposure to diethylstilbestrol (DES)
* current smoking > 10 cigarettes/day
* obesity-body mass index > 35
* history of clinical cardiovascular disease
* history of cerebrovascular disease
* history of thromboembolic disease
* coronary calcium score ≥ 50 units
* dyslipidemia-LDL cholesterol >190 mg/dl
* hypertriglyceridemia-triglycerides >400 mg/dl
* lipid lowering medication (statin, fibrate,or > 500 mg/day of niacin)
* nut allergy (Prometrium includes peanut oil)
* uncontrolled hypertension-systolic BP >150 and/or diastolic BP > 95
* hysterectomy
* history of, or prevalent, chronic diseases including any cancer (other than basal cell skin cancers), renal failure, cirrhosis, diabetes mellitus, and endocrinopathies other than adequately treated thyroid disease
* known HIV infection and/or medications for HIV infection
* results of any safety laboratory test chemistries, (TSH, CBC, U/A) more than 20% abnormal

Ages: 42 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 728 (Estimated)
Dates: Start 2005-09; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Rate of change of carotid intimal medial thickness by ultrasound | Measured at screening, 12, 24, 36, and 48 months

SECONDARY OUTCOMES:
Change in coronary calcium score by X-ray tomography | Meassured at screening and at 48 months
Plasma lipid profiles | Samples taken at screening , 12, 36, and 48 months
Blood clotting factors | Samples taken at screening, 12, 36 and 48 months
Serum inflammatory factors | Samples taken at screening, 12, 36 and 48 months
Hormone levels | Samples taken at screening, 12, 36 and 48 months
Cognitive and Affective scores on standard psychometric tests | Testing is conducted at Baseline, 18, 36 and 48 months
Quality of life | Measured at Baseline, 18, 36 and 48 months

CONTACTS AND LOCATIONS:
Overall Officials: S Mitchell Harman, MD, PhD, Study Director — Kronos Longevity Research Institute; Frederick Naftolin, MD, PhD, Study Director — Kronos Longevity Research Institute; Michael Mendelsohn, MD, Principal Investigator — Tufts Medical Center; Howard Hodis, MD, Principal Investigator — University of Southern California; Matthew Budoff, MD, Principal Investigator — University of California, Los Angeles; Sanjay Asthana, MD, Principal Investigator — University of Wisconsin, Madison; Dennis M Black, PhD, Principal Investigator — University of California, San Francisco
Locations (9):
- United States (9):
  - Kronos Longevity Research Institute, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - Yale University Medical Center, New Haven, Connecticut
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia Presbyterian Hospital, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - University of Utah, Salt Lake City, Utah
  - University of Washington/VA Puget Sound, HCS, Seattle/Tacoma, Washington

REFERENCES:
- [Background] Harman SM, Naftolin F, Brinton EA, Judelson DR. Is the estrogen controversy over? Deconstructing the Women's Health Initiative study: a critical evaluation of the evidence. Ann N Y Acad Sci. 2005 Jun;1052:43-56. doi: 10.1196/annals.1347.004. PMID 16024750
- [Background] Harman SM, Brinton EA, Cedars M, Lobo R, Manson JE, Merriam GR, Miller VM, Naftolin F, Santoro N. KEEPS: The Kronos Early Estrogen Prevention Study. Climacteric. 2005 Mar;8(1):3-12. doi: 10.1080/13697130500042417. PMID 15804727
- [Background] Harman SM, Brinton EA, Clarkson T, Heward CB, Hecht HS, Karas RH, Judelson DR, Naftolin F. Is the WHI relevant to HRT started in the perimenopause? Endocrine. 2004 Aug;24(3):195-202. doi: 10.1385/ENDO:24:3:195. PMID 15542885
- [Derived] Kara F, Tosakulwong N, Lesnick TG, Fought AJ, Kendell-Thomas J, Kapoor E, Faubion LL, Schwarz CG, Senjem ML, Fields JA, Min PH, Lowe VJ, Jack CR Jr, Bailey KR, James TT, Lobo RA, Manson JE, Pal L, Hammers DB, Malek-Ahmadi M, Cedars MI, Naftolin FN, Santoro N, Miller VM, Harman SM, Dowling NM, Gleason CE, Kantarci K. Associations of blood pressure with white matter hyperintensities later in life; influence of short-term menopausal hormone therapy. Menopause. 2025 Jan 1;32(1):12-22. doi: 10.1097/GME.0000000000002481. PMID 39729067
- [Derived] Kling JM, Dowling NM, Bimonte-Nelson H, Gleason CE, Kantarci K, Stonnington CM, Harman SM, Naftolin F, Pal L, Cedars M, Manson JE, James TT, Brinton EA, Miller VM. Associations between pituitary-ovarian hormones and cognition in recently menopausal women independent of type of hormone therapy. Maturitas. 2023 Jan;167:113-122. doi: 10.1016/j.maturitas.2022.10.002. Epub 2022 Oct 27. PMID 36395695
- [Derived] Kling JM, Miller VM, Tosakulwong N, Lesnick T, Kantarci K. Associations of pituitary-ovarian hormones and white matter hyperintensities in recently menopausal women using hormone therapy. Menopause. 2020 Aug;27(8):872-878. doi: 10.1097/GME.0000000000001557. PMID 32520900
- [Derived] El Khoudary SR, Venugopal V, Manson JE, Brooks MM, Santoro N, Black DM, Harman M, Naftolin F, Hodis HN, Brinton EA, Miller VM, Taylor HS, Budoff MJ. Heart fat and carotid artery atherosclerosis progression in recently menopausal women: impact of menopausal hormone therapy: The KEEPS trial. Menopause. 2020 Mar;27(3):255-262. doi: 10.1097/GME.0000000000001472. PMID 32015261
- [Derived] El Khoudary SR, Zhao Q, Venugopal V, Manson JE, Brooks MM, Santoro N, Black DM, Harman SM, Cedars MI, Hopkins PN, Kearns AE, Miller VM, Taylor HS, Budoff MJ. Effects of Hormone Therapy on Heart Fat and Coronary Artery Calcification Progression: Secondary Analysis From the KEEPS Trial. J Am Heart Assoc. 2019 Aug 6;8(15):e012763. doi: 10.1161/JAHA.119.012763. Epub 2019 Aug 1. PMID 31652073
- [Derived] Jayawardena E, Li D, Nakanishi R, Dey D, Dailing C, Qureshi A, Dickens B, Hathiramani N, Kim M, Flores F, Kearns AE, Lui LY, Black D, Budoff MJ. Non-contrast cardiac CT-based quantitative evaluation of epicardial and intra-thoracic fat in healthy, recently menopausal women: Reproducibility data from the Kronos Early Estrogen Prevention Study. J Cardiovasc Comput Tomogr. 2020 Jan-Feb;14(1):55-59. doi: 10.1016/j.jcct.2019.05.004. Epub 2019 May 4. PMID 31078511
- [Derived] Taylor HS, Tal A, Pal L, Li F, Black DM, Brinton EA, Budoff MJ, Cedars MI, Du W, Hodis HN, Lobo RA, Manson JE, Merriam GR, Miller VM, Naftolin F, Neal-Perry G, Santoro NF, Harman SM. Effects of Oral vs Transdermal Estrogen Therapy on Sexual Function in Early Postmenopause: Ancillary Study of the Kronos Early Estrogen Prevention Study (KEEPS). JAMA Intern Med. 2017 Oct 1;177(10):1471-1479. doi: 10.1001/jamainternmed.2017.3877. PMID 28846767
- [Derived] Cintron D, Beckman JP, Bailey KR, Lahr BD, Jayachandran M, Miller VM. Plasma orexin A levels in recently menopausal women during and 3 years following use of hormone therapy. Maturitas. 2017 May;99:59-65. doi: 10.1016/j.maturitas.2017.01.016. Epub 2017 Feb 17. PMID 28364870
- [Derived] Owen CM, Pal L, Mumford SL, Freeman R, Isaac B, McDonald L, Santoro N, Taylor HS, Wolff EF. Effects of hormones on skin wrinkles and rigidity vary by race/ethnicity: four-year follow-up from the ancillary skin study of the Kronos Early Estrogen Prevention Study. Fertil Steril. 2016 Oct;106(5):1170-1175.e3. doi: 10.1016/j.fertnstert.2016.06.023. Epub 2016 Jul 5. PMID 27393520
- [Derived] Gleason CE, Dowling NM, Wharton W, Manson JE, Miller VM, Atwood CS, Brinton EA, Cedars MI, Lobo RA, Merriam GR, Neal-Perry G, Santoro NF, Taylor HS, Black DM, Budoff MJ, Hodis HN, Naftolin F, Harman SM, Asthana S. Effects of Hormone Therapy on Cognition and Mood in Recently Postmenopausal Women: Findings from the Randomized, Controlled KEEPS-Cognitive and Affective Study. PLoS Med. 2015 Jun 2;12(6):e1001833; discussion e1001833. doi: 10.1371/journal.pmed.1001833. eCollection 2015 Jun. PMID 26035291
- [Derived] Harman SM, Black DM, Naftolin F, Brinton EA, Budoff MJ, Cedars MI, Hopkins PN, Lobo RA, Manson JE, Merriam GR, Miller VM, Neal-Perry G, Santoro N, Taylor HS, Vittinghoff E, Yan M, Hodis HN. Arterial imaging outcomes and cardiovascular risk factors in recently menopausal women: a randomized trial. Ann Intern Med. 2014 Aug 19;161(4):249-60. doi: 10.7326/M14-0353. PMID 25069991
- [Derived] Dowling NM, Gleason CE, Manson JE, Hodis HN, Miller VM, Brinton EA, Neal-Perry G, Santoro MN, Cedars M, Lobo R, Merriam GR, Wharton W, Naftolin F, Taylor H, Harman SM, Asthana S. Characterization of vascular disease risk in postmenopausal women and its association with cognitive performance. PLoS One. 2013 Jul 17;8(7):e68741. doi: 10.1371/journal.pone.0068741. Print 2013. PMID 23874743
- [Derived] Ogorodnikova AD, Khan UI, McGinn AP, Zeb I, Budoff MJ, Harman SM, Miller VM, Brinton EA, Manson JE, Hodis HN, Merriam GR, Cedars MI, Taylor HS, Naftolin F, Lobo RA, Santoro N, Wildman RP. Ectopic fat and adipokines in metabolically benign overweight/obese women: the Kronos Early Estrogen Prevention Study. Obesity (Silver Spring). 2013 Aug;21(8):1726-33. doi: 10.1002/oby.20200. Epub 2013 May 13. PMID 23670850
- [Derived] Farr JN, Khosla S, Miyabara Y, Miller VM, Kearns AE. Effects of estrogen with micronized progesterone on cortical and trabecular bone mass and microstructure in recently postmenopausal women. J Clin Endocrinol Metab. 2013 Feb;98(2):E249-57. doi: 10.1210/jc.2012-3406. Epub 2013 Jan 15. PMID 23322818
- [Derived] Wolff EF, He Y, Black DM, Brinton EA, Budoff MJ, Cedars MI, Hodis HN, Lobo RA, Manson JE, Merriam GR, Miller VM, Naftolin F, Pal L, Santoro N, Zhang H, Harman SM, Taylor HS. Self-reported menopausal symptoms, coronary artery calcification, and carotid intima-media thickness in recently menopausal women screened for the Kronos early estrogen prevention study (KEEPS). Fertil Steril. 2013 Apr;99(5):1385-91. doi: 10.1016/j.fertnstert.2012.11.053. Epub 2013 Jan 8. PMID 23312232
- [Derived] Huang G, Wang D, Khan UI, Zeb I, Manson JE, Miller V, Hodis HN, Budoff MJ, Merriam GR, Harman MS, Brinton EA, Cedars MI, Su Y, Lobo RA, Naftolin F, Santoro N, Taylor HS, Wildman RP. Associations between retinol-binding protein 4 and cardiometabolic risk factors and subclinical atherosclerosis in recently postmenopausal women: cross-sectional analyses from the KEEPS study. Cardiovasc Diabetol. 2012 May 15;11:52. doi: 10.1186/1475-2840-11-52. PMID 22587616
- [Derived] Huang G, Wang D, Zeb I, Budoff MJ, Harman SM, Miller V, Brinton EA, El Khoudary SR, Manson JE, Sowers MR, Hodis HN, Merriam GR, Cedars MI, Taylor HS, Naftolin F, Lobo RA, Santoro N, Wildman RP. Intra-thoracic fat, cardiometabolic risk factors, and subclinical cardiovascular disease in healthy, recently menopausal women screened for the Kronos Early Estrogen Prevention Study (KEEPS). Atherosclerosis. 2012 Mar;221(1):198-205. doi: 10.1016/j.atherosclerosis.2011.12.004. Epub 2011 Dec 9. PMID 22209479
- [Derived] Henderson VW. Aging, estrogens, and episodic memory in women. Cogn Behav Neurol. 2009 Dec;22(4):205-14. doi: 10.1097/WNN.0b013e3181a74ce7. PMID 19996872
- [Derived] Mulvagh SL, Behrenbeck T, Lahr BA, Bailey KR, Zais TG, Araoz PA, Miller VM. Endothelial function and cardiovascular risk stratification in menopausal women. Climacteric. 2010 Feb;13(1):45-54. doi: 10.3109/13697130902943287. PMID 19657788
- See also: Information on hormone treatment and KEEPS rationale — http://www.keepstudy.org
- See also: Information on sponsoring institution — http://www.kronosinstitute.org